CLINICAL TRIAL: NCT01592253
Title: Investigation of the Safety and Immunologic Biomarker After Conversion From Calcineurin Inhibitor to Rapamune in Stable Renal Transplant Recipient
Brief Title: Study to Evaluate Safety and Immunologic Biomarker of Rapamune in Patients With Stable Renal Transplant Recipient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, ChulWoo Yang, professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RAPA CONVERT TRIAL
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Acute Rejection of Renal Transplant
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sirolimus — Beginning on day, an initial maintenance dose of 2mg/day should be given. A trough level should be obtained between days 3 and 8, and the daily dose of sirolimus should be adjusted thereafter.

SUMMARY:
For patients who meet the inclusion criteria and who agree to participate in this study, the investigators sampled peripheral blood 10cc and performed the analysis for immunologic profile just before the conversion of immune suppressant. At 1 month, 6 month, and 1 year from the conversion of Immune suppressant (CNI to rapamune), the investigators performed tha analysis fo immune profile again. During the study period, the interval of the visit of subclinic and the kinds of laboratory test (Blood and urine test) would not change compared to before the start of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant recipient who has passed at least 10 years
2. No acute rejection episode during the previous 6 months
3. No change of prescription of immune suppressants
4. Normal allograft function (MDRD eGFR > 80 mL/min/1.73 m2)
5. Change of allograft function less than 10 % of baseline value durant the previous 1 year
6. No proteinuria and hematuria

Exclusion Criteria:

1. Patients who donut want to participate in this study
2. Patients who should continue immune suppressant due to another cause (e/g combined autoimmune disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
biopsy proven acute rejection | Study duration is 12 months
  Number of episode of biopsy proven acute rejection

SECONDARY OUTCOMES:
Serum Creatinine, MDRD eGFR | Study duration is 12 months
  Mean diurnal Serum Creatinine, MDRD eGFR change of greater than or equal to 20% at month 12 vs baseline

CONTACTS AND LOCATIONS:
Overall Officials: ChulWoo Yang, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul, South Korea